CLINICAL TRIAL: NCT04098913
Title: The Short Term Efficacy of Reducing Screen-based Media Use on Physical Activity, Sleep, and Physiological Stress and Well-Being in Families With Children - A Randomized Controlled Trial
Brief Title: Short-term Efficacy of Reducing Screen-based Media Use
Acronym: SCREENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: European Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20170213 (2)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Screen Time
Keywords: screen time; physical activity; sleep; stress
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced screen-based media use (Experimental): Reducing recreational screen-based media use for a period of 2 weeks.
  Interventions: Behavioral: Reduced screen-based media use
- Control group (No Intervention): Participants are asked to continue their habitual screen-based media use.

INTERVENTIONS:
Behavioral: Reduced screen-based media use — Participants must remove all recreational screen-based media use beyond 3 hours/week. This includes all recreational screen-based media use inside and outside the household. As a tool to comply with the intervention the families will hand-over all portable screen-based media devices. In return, each participant who own a smartphone will receive a regular cell-phone which can only make phone calls and send text messages. For a maximum of ½ an hour a day, adult participants may use screen-based media for necessary contact/errands. If one of the adult participants can not hand over their smartphones due to daily use for work purposes we will install an app tracking screen use on these devices.
  Arms: Reduced screen-based media use

SUMMARY:
The purpose of this randomized controlled trial is to investigate the short-term efficacy of reducing recreational screen-based media use on physical activity patterns, sleep, physiological stress in families at least one child between 6-10 years of age.

DETAILED DESCRIPTION:
Today screen-based media devices are almost unavoidable in our everyday lives. The media landscape has changed markedly during the past decade with some of the main aspects being the introduction of new portable devices, social networks, and online streaming services. The current experimental evidence on the efficacy of reducing todays screen-based media use in free-living is scarce.

This randomized controlled trial will be carried out based on the experience from a recently conducted pilot study, which was a 2-arm randomized non-controlled trial. The purposes of the pilot study were to explore the feasibility of our recruitment protocol, 7-day measurement protocol and the degree of compliance to the intervention components; namely a heavy restriction in recreational screen time for a 2-week period, either timed (no screen after 18 pm) or time restricted (≤ 3 hours/week/person).

In the current trial, only the time restricted protocol will be included, compared to a control group. To investigate the short-term efficacy of the intervention, the participants will go through a 7-day measurement protocol at baseline and again, during the final week of the intervention period (follow-up).

Ninety-five families with at least one child between 6-10 years of age will be recruited. A randomly selected adult from each household will be invited to answer a questionnaire, also including an invitation regarding participation in the current randomized controlled trial. Invitations will be sent to the adults' digital mailbox (e-boks), which is an online solution where one can receive mail from e.g. Danish public authorities. Based on the answers in the survey a preliminary screening for eligibility will be conducted (see section on inclusion/exclusion criteria). Families who fulfill specific criteria in the survey and further criteria assessed during a phone conversation will be invited to participate in this randomized controlled trial. Families who wish to participate will, after completion of the baseline protocol, will be randomized to either the intervention group or the control group (see section on arms and interventions).

The intervention (reducing recreational screen-based media use) was designed using the core major and minor elements of Albert Bandura's Social Cognitive Theory; namely, based on the idea of reciprocal determinism of an individual's environment, personal factors and behavior. The intervention includes i) a preparation document and meeting with the parents with the purpose of planning the course of the intervention and prepare the parents to set goals and self-regulate; ii) handing over the families portable screen devices when possible with an alternative mobile phone in exchange, which can be solely used for calls and text messages, will be afforded to the participants; iii) installing monitor software on all computers (stationary and laptops) and tablets and smartphone if these could not be given up, and connect a monitor device to all televisions in each household; iv) using "intervention reminders" (social cues), which will be placed beside stationary screen-based media devices and at central positions in the household such as the dining table.

ELIGIBILITY:
Inclusion Criteria:

* High amount of screen time according to self-report: In each household, at least one adult must be above the 40th percentile for self-reported screen-time during spare time based on what was reported in the survey ((characterized as high in this study).
* To be eligible for the measurements children in the household must be ≥ 4 and < 15 years old during the entire experiment period.
* Adults must work full time or be full-time students
* Adults and children who participates in the measurements must have the resources to remove all recreational- and work-/school-related screen-time in the late afternoon and evening hours and during weekend days, with a few exceptions (described in the "intervention" section below), for a period of 2 weeks (intervention length).
* The household must include at least one adult and one child 6-10 years of age at the time the survey was sent out, both of whom must consent to participate in the experiment.
* Participants must report that they consider the extent of their screen time an issue
* Participants must report to be particularly motivated to decrease screen-time for the whole family household.
* Members of the household who choose not to participate or who is ineligible to participate in the measurements or the intervention, must be willing to support the remainder of the household in making the experiment a success for them.

Exclusion Criteria:

* If the adults or children only reside in the household part time, e.g. have multiple addresses
* Prescribed a period of sick leave due to stress within the last 3 months.
* Diagnosis of sleep disorders from their general practitioner still interfering sleep
* Working night shifts
* In any shape or form limited in one's ability to engage in physical activities
* Neuro psychiatric disorders, such as attention deficit hyperactivity disorder (ADHD) and autism

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Between group change in leisure time spent being non-sedentary (children) | 14 days (experiment period)
  Non-sedentary time is defined as any waking activity characterized as not being in a sitting, reclining or lying posture with minimal stationary movement. Activity is measured for 7 consecutive days at baseline and follow-up using combined trunk- and thigh worn accelerometry (Axivity AX3).

SECONDARY OUTCOMES:
Between group change in leisure time spent being non-sedentary(adults) | 14 days (experiment period)
  Non-sedentary time is defined as any waking activity characterized as not being in a sitting, reclining or lying posture with minimal stationary movement. Activity is measured for 7 consecutive days at baseline and follow-up using combined trunk- and thigh worn accelerometry (Axivity AX3).
Between group change in leisure time moderate to vigorous physical activity (MVPA) (children) | 14 days (experiment period)
  Activity is measured for 7 consecutive days at baseline and follow-up using combined trunk- and thigh worn accelerometry (Axivity AX3).
Between group change in leisure time moderate to vigorous physical activity MVPA (adults) | 14 days (experiment period)
  Activity is measured for 7 consecutive days at baseline and follow-up using combined trunk- and thigh worn accelerometry (Axivity AX3).
Between group change in leisure time spent being non-sedentary on weekdays (children) | 14 days (experiment period)
  Non-sedentary time is defined as any waking activity characterized as not being in a sitting, reclining or lying posture with minimal stationary movement. Activity is measured for 7 consecutive days at baseline and follow-up using combined trunk- and thigh worn accelerometry (Axivity AX3).
Between group change in leisure time spent being non-sedentary on weekdays (adults) | 14 days (experiment period)
  Non-sedentary time is defined as any waking activity characterized as not being in a sitting, reclining or lying posture with minimal stationary movement. Activity is measured for 7 consecutive days at baseline and follow-up using combined trunk- and thigh worn accelerometry (Axivity AX3).
Between group change in leisure time spent being non-sedentary on weekend days (children) | 14 days (experiment period)
  Non-sedentary time is defined as any waking activity characterized as not being in a sitting, reclining or lying posture with minimal stationary movement. Activity is measured for 7 consecutive days at baseline and follow-up using combined trunk- and thigh worn accelerometry (Axivity AX3).
Between group change in leisure time spent being non-sedentary on weekend days (adults) | 14 days (experiment period)
  Non-sedentary time is defined as any waking activity characterized as not being in a sitting, reclining or lying posture with minimal stationary movement. Activity is measured for 7 consecutive days at baseline and follow-up using combined trunk- and thigh worn accelerometry (Axivity AX3).
Between group change in total sleep duration (children) | 14 days (experiment period)
  Total sleep duration is defined as time spent asleep within a sleep period, excluding wake time. Total sleep duration is measured for three consecutive nights at baseline and follow-up using single channel EEG-based sleep equipment (Zmachine insight+).
Between group change in total sleep duration (adults) | 14 days (experiment period)
  Total sleep duration is defined as time spent asleep within a sleep period, excluding wake time. Total sleep duration is measured for three consecutive nights at baseline and follow-up using single channel EEG-based sleep equipment (Zmachine insight+).
Between group change in sleep onset latency (children) | 14 days (experiment period)
  Sleep is measured for three consecutive nights at baseline and follow-up using single channel EEG-based sleep equipment (Zmachine insight+). Sleep onset latency is calculated using the EEG-based sleep stages.
Between group change in sleep onset latency (adults) | 14 days (experiment period)
  Sleep is measured for three consecutive nights at baseline and follow-up using single channel EEG-based sleep equipment (Zmachine insight+). Sleep onset latency is calculated using the EEG-based sleep stages.
Between group change in wake after sleep onset (children) | 14 days (experiment period)
  Sleep is measured for three consecutive nights at baseline and follow-up using single channel EEG-based sleep equipment (Zmachine insight+). Wake after sleep onset is calculated using the EEG-based sleep stages.
Between group change in wake after sleep onset (adults) | 14 days (experiment period)
  Sleep is measured for three consecutive nights at baseline and follow-up using single channel EEG-based sleep equipment (Zmachine insight+). Wake after sleep onset is calculated using the EEG-based sleep stages.
Between group change in sleep stages (awake, light sleep, deep sleep, REM-sleep) (children) | 14 days (experiment period)
  Sleep stages are measured for three consecutive nights at baseline and follow-up using single channel EEG-based sleep equipment (Zmachine insight+).
Between group change in sleep stages (awake, light sleep, deep sleep, REM-sleep) (adults) | 14 days (experiment period)
  Sleep stages are measured for three consecutive nights at baseline and follow-up using single channel EEG-based sleep equipment (Zmachine insight+).

OTHER OUTCOMES:
Between group change in cortisol awakening response (adults) | 14 days (experiment period)
  Cortisol awakening response is measured using saliva samples. Samples are collected at awakening, 30 minutes after awakening, and 45 minutes after awakening for three consecutive days.
Between group change in diurnal cortisol slope (adults) | 14 days (experiment period)
  The diurnal cortisol slope is measured using saliva samples. Samples are collected at bedtime and immediate after awakening, and the diurnal cortisol slope will be calculated as the difference in waking and bedtime cortisol levels summarized based on assessments over three consecutive days.
Between group change in heart rate variability (HRV) | 14 days (experiment period)
  Heart Rate Variability is recorded for 72 consecutive hours at baseline and follow-up using Firstbeat 2 (time- and frequency domain measures).
Between group change in non-metabolic heart rate variability (adults) | 14 days (experiment period)
  Heart Rate Variability is recorded for 72 consecutive hours at baseline and follow-up using Firstbeat 2. Non-metabolic heart rate variability is quantified by removing the effect of physical activity.
Between group change in mood disturbance score (adults) | 14 days (experiment period)
  Mood states are assessed using the Profile of moods, which is a 65-item questionnaire each item is scored from 0-4. The questionnaire is divided into 6 subscales 1) Tension, 2) Depression, 3) Anger, 4) Fatigue, 5) Confusion, and 6) Vigour. High vigour score represents good mood and low scores on the other subscales represent good mood. The total mood disturbance score is calculated by adding subscales 1-5 and subtracting subscale 6.
Between group change in WHO-5-score (adults) | 14 days (experiment period)
  WHO-5 is a questionnaire measuring current mental well-being. The questionnaire consist of 5 item each scores from 0-5. Scores from each item are added and multiplied by 4. This results in a score between 0-100, lower scores indicate lower mental well-being.
Between group change in the total difficulties score (children) | 14 days (experiment period)
  The strengths and difficulties questionnaire (SDQ) is divided into 5 subscales 1) emotional symptoms scale, 2) conduct problem scale, 3) hyperactivity scale, 4) peer problem scale, and 5) prosocial scale. The subscales are scored from 0-10. Lower scores indicate low difficulties on subscale 1-4. Lower scores indicate low amount of social strengths on subscale 5. The total difficulties score will be calculated from the summary scores from subscale 1-4.
Between group change in subjective sleep quality (adults) | 14 days (experiment period)
  Quality of sleep is assessed using the quality of sleep subscale (item 4-5) from the Leeds Sleep Evaluation Questionnaire. Each item consist of a visual analog scale (0-100), where lower scores = higher symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Grøntved, Ph.D., Principal Investigator — University of Southern Denamrk
Locations (1):
- University of Southern Denmark, Odense, Funen, Denmark

REFERENCES:
- [Derived] Schmidt-Persson J, Rasmussen MGB, Sorensen SO, Mortensen SR, Olesen LG, Brage S, Kristensen PL, Bilenberg N, Grontved A. Screen Media Use and Mental Health of Children and Adolescents: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2419881. doi: 10.1001/jamanetworkopen.2024.19881. PMID 38995646
- [Derived] Pedersen J, Rasmussen MGB, Sorensen SO, Mortensen SR, Olesen LG, Brage S, Kristensen PL, Puterman E, Grontved A. Effects of limiting digital screen use on well-being, mood, and biomarkers of stress in adults. Npj Ment Health Res. 2022;1(1):14. doi: 10.1038/s44184-022-00015-6. Epub 2022 Oct 12. PMID 37521498
- [Derived] Pedersen J, Rasmussen MGB, Sorensen SO, Mortensen SR, Olesen LG, Brond JC, Brage S, Kristensen PL, Grontved A. Effects of Limiting Recreational Screen Media Use on Physical Activity and Sleep in Families With Children: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2022 Aug 1;176(8):741-749. doi: 10.1001/jamapediatrics.2022.1519. PMID 35604678
- [Derived] Rasmussen MGB, Pedersen J, Olesen LG, Brage S, Klakk H, Kristensen PL, Brond JC, Grontved A. Short-term efficacy of reducing screen media use on physical activity, sleep, and physiological stress in families with children aged 4-14: study protocol for the SCREENS randomized controlled trial. BMC Public Health. 2020 Mar 23;20(1):380. doi: 10.1186/s12889-020-8458-6. PMID 32293374

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT04098913/SAP_000.pdf